CLINICAL TRIAL: NCT06197243
Title: Augmenting Benzodiazepine Receptor Agonist Deprescribing With Acupuncture and Yoga
Brief Title: Augmenting Benzodiazepine Receptor Agonist Deprescribing With Acupuncture and Yoga Among Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Gurjeet Birdee, Director, Osher Center for Integrative Health Department of Physical Medicine and Rehabilitation, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 230716; R24AG064025 (NIH)
Record Dates: First submitted 2023-12-26; First posted 2024-01-09 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-05

CONDITIONS: Anxiety; Insomnia; Benzodiazepine; Deprescription
MeSH Terms: conditions — Anxiety Disorders; Sleep Initiation and Maintenance Disorders | interventions — Acupuncture Therapy; Yoga; Deprescriptions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Feasibility, Adherence and Acceptability Measure (Experimental): Assay of feasibility of study enrollment and feasibility of study treatments, the latter of which is measured via fidelity, adherence, and acceptability of/to treatments and interventions. Interventions administered for 12 weeks. Fidelity, adherence, and acceptability will be measured via patient survey and engagement.
  Interventions: Other: Acupuncture; Other: Yoga; Other: Deprescribing

INTERVENTIONS:
Other: Acupuncture — Patients will receive acupuncture for 12 weeks.
Other: Yoga — Patients will receive yoga therapy with one of three yoga instructors. Patients will remain with singular yoga instructor for duration of study. It is anticipated that patients will participate in yoga therapy for 12 weeks at home and in-clinic.
Other: Deprescribing — Deprescribing of patients' benzodiazepine use will be monitored by psychiatric nurse. Tapering method will be followed for medication deprescription.

SUMMARY:
The main purpose of this 12-week study is to see if a new combination of treatments can help older adults reduce benzodiazepine or related medication use. The treatment combination consists of 1) medical provider visits to gradually reduce the medication dose over 12 weeks, 2) acupuncture treatments, and 3) private yoga classes. Participants will be offered weekly visits for 12 weeks to receive combined treatments. Participants will be provided surveys before, during, and after the study to learn about their experience of the treatments. At the end of the study, participants will be invited to participate in a focus group to learn about their experience in the study.

DETAILED DESCRIPTION:
This study consists of a single-arm clinical study among 30 older adults taking benzodiazepine receptor antagonists (BRZA) to assess the feasibility of protocol-driven BRZA deprescribing augmented with combined acupuncture and yoga. Adults 65 years or older that are taking BRZA will be recruited. Deprescribing will be provided at weekly visits with a psychiatric nurse practitioner at the Osher Center for Integrative Health at Vanderbilt University Medical Center. Participants will receive acupuncture and yoga from a staff acupuncturist and yoga instruction from a yoga instructor at the Osher Center. Feasibility of study enrollment will occur through the study enrollment period. Feasibility of study treatments will be evaluated during and after study treatment delivery. Feasibility of study outcome assessments will occur at baseline, 4, 8, and 12 weeks. Throughout the research process, investigators will engage a Stakeholder Advisory Panel consisting of patients and clinicians.

ELIGIBILITY:
Inclusion Criteria:

* 65 years and older
* Taking benzodiazepines or related medications (i.e. zolpidem, zopiclone, eszopiclone, zaleplon) at least 4 times in the last month
* English speaking
* Ability to understand study procedures and to comply with them for the length of the study

Exclusion Criteria:

* Cognitive impairment
* Drinking more than 3 alcoholic beverages per day
* Substance abuse disorder
* Uncontrolled psychiatric disorder, such as major depression or psychosis
* Inability or unwillingness of individual or legal guardian.representative to give written informed consent.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 23 (Actual)
Dates: Start 2023-12-14 (Actual); Primary Completion 2025-05-23 (Actual); Study Completion 2025-05-23 (Actual)

PRIMARY OUTCOMES:
BRZA dose change | Baseline to 12 weeks
  Dose of BRZA for patients will be measured at baseline, 4, 8, and 12 weeks

SECONDARY OUTCOMES:
Insomnia | Baseline to12 weeks
  Will use Patient Reported Outcomes Measurement Information System(PROMIS) Sleep Disturbance Computerized Adaptive Testing to assess difficulties staying and falling asleep. The minimum value is 0 and the maximum value is 100, with higher scores determining worse outcomes.
Anxiety | Baseline to 12 weeks
  Will use Patient Reported Outcomes Measurement Information System(PROMIS) Anxiety Computerized Adaptive Testing. The minimum value is 0 and the maximum value is 100, with higher scores determining worse outcomes.
Proportion of participants whom the investigators collect primary and secondary outcomes. | Baseline to 12 weeks
  Will estimate feasibility of data collection for study measures by calculating proportion of participants whom the investigators collect primary and secondary outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Gurjeet Birdee, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Osher Center for Integrative Health at Vanderbilt, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-07-09): https://cdn.clinicaltrials.gov/large-docs/43/NCT06197243/ICF_000.pdf